CLINICAL TRIAL: NCT01306929
Title: A Multi-Center, North American, Open-Label Extension Study of Pridopidine (ACR16) in the Symptomatic Treatment of Huntington's Disease (Open-HART).
Brief Title: Open-label Extension Study of Pridopidine (ACR16) in the Symptomatic Treatment of Huntington Disease
Acronym: OPEN-HART
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prilenia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACR16C015
Record Dates: First submitted 2011-02-28; First posted 2011-03-02 (Estimated); Results first posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Huntington Disease
Keywords: Huntington Disease.
MeSH Terms: conditions — Huntington Disease | interventions — pridopidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- pridopidine (Experimental): 45mg bid
  Interventions: Drug: pridopidine

INTERVENTIONS:
Drug: pridopidine — 45mg bid

SUMMARY:
Huntington disease (HD) is a hereditary neurodegenerative disorder causing impairment in movement, behavioral dysfunction and dementia. The movement disorder is mainly characterized by chorea (involuntary movements) and a progressive loss of voluntary movement causing a substantial functional impairment over time. The study will assess the long-term safety of pridopidine and the treatment effects during long-term, open-label treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to, and has provided written Informed Consent prior to any study related procedure.
* Patient has completed the HART (ACR16C009) or the PRIDE-HD (TV7820- CNS-20002) studies and had remained on IMP during the full on-treatment part of the study (including de-escalated patients) or has transitioned from the Open-HART pre-virtualization study period.
* Willing and able to take oral medication and able to comply with the study specific procedures.
* Patient has a wireless internet connection at home (and/or applicable locations) at the first remote visit.
* Patient has the ability to transition from in-person study visits to virtual study visits. The first remote visit (RV1) will take place within approximately 30 days after the last in-person visit.

  * Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* Ongoing treatment with tetrabenazine or deutetrabenazine, seizure threshold lowering medications, or certain antipsychotics and antidepressants.
* Newly instigated or changed treatment with neuroleptics/antipsychotics
* Use of tricyclic antidepressants or class I & III antiarrhythmics at any time during the study period.
* Severe intercurrent illness that, in the opinion of the Investigator (or qualified designee), may put the subject at risk when continuing participation in the study.
* Alcohol and/or drug abuse as defined by the Diagnostic and Statistical Manual - Fourth Edition - Text Revision criteria for substance abuse - this includes the illicit use of cannabis.
* Subjects with a known history of epilepsy or a history of febrile seizure(s) or seizure(s) of unknown cause.
* Females who are pregnant or lactating.
* Females who are of child bearing potential and not taking adequate contraceptive precautions (either oral, barrier or chemical contraceptives) are excluded from the trial. Females of child bearing potential taking acceptable contraceptive precautions can be included.
* Known allergy to any ingredients of the trial medication.

  * Additional criteria apply, please contact the investigator for more information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2011-03-24 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2018-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: See Central Contact section for questions about, Principal Investigator — study officials

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McGarry A, Auinger P, Kieburtz K, Geva M, Mehra M, Abler V, Grachev ID, Gordon MF, Savola JM, Gandhi S, Papapetropoulos S, Hayden M. Additional Safety and Exploratory Efficacy Data at 48 and 60 Months from Open-HART, an Open-Label Extension Study of Pridopidine in Huntington Disease. J Huntingtons Dis. 2020;9(2):173-184. doi: 10.3233/JHD-190393. PMID 32508327
- [Derived] McGarry A, Kieburtz K, Abler V, Grachev ID, Gandhi S, Auinger P, Papapetropoulos S, Hayden M. Safety and Exploratory Efficacy at 36 Months in Open-HART, an Open-Label Extension Study of Pridopidine in Huntington's Disease. J Huntingtons Dis. 2017;6(3):189-199. doi: 10.3233/JHD-170241. PMID 28826192

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited adult patients with Huntington's Disease (HD) who had completed studies ACR16C009 (NCT00724048) or TV7820-CNS-20002 (NCT02006472). The first patient was recruited on 24 Mar 2011, and the last patient completed the trial on 5 Jan 2018.
Groups:
- Pridopidine: Pridopidine 45 mg twice daily (bid), taken once in the morning and once in the afternoon.
Period: Overall Study
Arm/Group | Pridopidine
Started | 134
Completed | 40
Not Completed | 94
Not completed — Withdrawal by Subject | 23
Not completed — Adverse Event | 21
Not completed — Physician Decision | 13
Not completed — Death | 8
Not completed — Withdrawal by parent/guardian | 5
Not completed — Protocol Violation | 3
Not completed — Non-compliance with study drug | 2
Not completed — Lost to Follow-up | 2
Not completed — Various | 17

BASELINE CHARACTERISTICS:
Arm/Group | Pridopidine
Number analyzed (Participants) | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 129
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  Canada | 50
  United States | 84
Weight [Mean (Standard Deviation); unit: kg] — Population: Data available for 132 of 134 patients.
  kg
    number analyzed (Participants) | 132
    (all) | 74.7 (18.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With at Least One Adverse Event
Time Frame: From signing of the informed consent through the end of the follow-up period, which was defined as 30 days after the final study visit in an individual patient, an average of 2.8 years
Population: Safety analysis set, including all enrolled patients who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pridopidine
Number analyzed (Participants) | 134
Participants | 119

2. Secondary Outcome: Unified Huntington's Disease Rating Scale (UHDRS) Total Motor Score (TMS)
Description: TMS was defined as the sum of all UHDRS motor domains ratings. The motor section of the UHDRS assesses motor features of Huntington's Disease (HD) with standardized ratings of oculo-motor function, dysarthria, chorea, dystonia, gait, and postural stability. Each of 31 assessments is rated on a scale of 0 (normal) to 4 (marked impairment) for a TMS range of 0-124.
Time Frame: Baseline and at Month 12, 24, 36, 48, 60, and 72
Population: Full analysis set, comprising all enrolled patients who received at least 1 dose of study drug and had a baseline and at least 1 post-baseline UHDRS-TMS assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pridopidine
Number analyzed (Participants) | 123
score on a scale
  Baseline | 38.3 (15.2)
  Month 12: number analyzed (Participants) | 118
  Month 12 | 41.5 (18.7)
  Month 24: number analyzed (Participants) | 74
  Month 24 | 41.7 (20.7)
  Month 36: number analyzed (Participants) | 59
  Month 36 | 44.7 (19.8)
  Month 48: number analyzed (Participants) | 49
  Month 48 | 45.3 (19.7)
  Month 60: number analyzed (Participants) | 35
  Month 60 | 45.7 (20.6)
  Month 72: number analyzed (Participants) | 30
  Month 72 | 50.0 (23.2)

ADVERSE EVENTS:
Time Frame: From signing of the informed consent through the end of the follow-up period, which was defined as 30 days after the final study visit in an individual patient, an average of 2.8 years
Arm/Group | Pridopidine
All-Cause Mortality (participants affected / at risk) | 8/134
Serious Adverse Events (participants affected / at risk) | 31/134
Other Adverse Events (participants affected / at risk) | 119/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pridopidine (N=134)
Arteriosclerosis cornonary artery (Cardiac disorders) | 1 (1)
Bungle branch block right (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (5)
Subdural haematoma (Injury, poisoning and procedural complications) | 4 (5)
Skull fracture (Injury, poisoning and procedural complications) | 2 (2)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Starvation (Metabolism and nutrition disorders) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Convulsion (Nervous system disorders) | 2 (3)
Loss of consciousness (Nervous system disorders) | 2 (2)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2)
Balance disorder (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Encephalitis (Nervous system disorders) | 1 (1)
Status migrainosus (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Intentional self-injury (Psychiatric disorders) | 2 (2)
Abnormal behaviour (Psychiatric disorders) | 1 (1)
Aggression (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pridopidine (N=134)
Anaemia (Blood and lymphatic system disorders) | 6 (6)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2)
Aortic valve incompetence (Cardiac disorders) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (2)
Bradycardia (Cardiac disorders) | 1 (1)
Bundle branch block right (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (3)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1)
Asthenopia (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (2)
Conjunctival haemorrhage (Eye disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Macular degeneration (Eye disorders) | 1 (1)
Photopsia (Eye disorders) | 1 (1)
Retinal tear (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 16 (19)
Nausea (Gastrointestinal disorders) | 11 (15)
Vomiting (Gastrointestinal disorders) | 10 (17)
Constipation (Gastrointestinal disorders) | 7 (7)
Dysphagia (Gastrointestinal disorders) | 7 (8)
Dry mouth (Gastrointestinal disorders) | 5 (5)
Dental caries (Gastrointestinal disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 4 (4)
Faecal incontinence (Gastrointestinal disorders) | 4 (4)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Colitis ulcerative (Gastrointestinal disorders) | 2 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (3)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gingival disorder (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Periodontitis (Gastrointestinal disorders) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Tongue disorder (Gastrointestinal disorders) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 1 (1)
Irritability (General disorders) | 13 (17)
Gait disturbance (General disorders) | 8 (9)
Fatigue (General disorders) | 4 (4)
Pyrexia (General disorders) | 4 (4)
Asthenia (General disorders) | 3 (3)
Cyst (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 2 (4)
Chest pain (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (2)
Nasopharyngitis (Infections and infestations) | 16 (22)
Upper respiratory tract infection (Infections and infestations) | 9 (17)
Sinusitis (Infections and infestations) | 8 (11)
Urinary tract infection (Infections and infestations) | 8 (19)
Bronchitis (Infections and infestations) | 7 (7)
Influenza (Infections and infestations) | 6 (9)
Gastroenteritis (Infections and infestations) | 4 (4)
Ear infection (Infections and infestations) | 3 (3)
Tooth abscess (Infections and infestations) | 3 (3)
Clostridium difficile colitis (Infections and infestations) | 2 (3)
Fungal skin infection (Infections and infestations) | 2 (2)
Furuncle (Infections and infestations) | 2 (2)
Herpes zoster (Infections and infestations) | 2 (2)
Hordeolum (Infections and infestations) | 2 (2)
Onychomycosis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (4)
Diverticulitis (Infections and infestations) | 1 (1)
Enterococcal infection (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Gingival infection (Infections and infestations) | 1 (1)
Infected dermal cyst (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Oral fungal infection (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 46 (148)
Contusion (Injury, poisoning and procedural complications) | 18 (28)
Laceration (Injury, poisoning and procedural complications) | 18 (32)
Excoriation (Injury, poisoning and procedural complications) | 11 (15)
Accidental overdose (Injury, poisoning and procedural complications) | 3 (3)
Head injury (Injury, poisoning and procedural complications) | 3 (4)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3)
Muscle strain (Injury, poisoning and procedural complications) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3)
Rib fracture (Injury, poisoning and procedural complications) | 3 (3)
Arthropod sting (Injury, poisoning and procedural complications) | 2 (2)
Clavicle fracture (Injury, poisoning and procedural complications) | 2 (3)
Facial bones fracture (Injury, poisoning and procedural complications) | 2 (2)
Lip injury (Injury, poisoning and procedural complications) | 2 (3)
Overdose (Injury, poisoning and procedural complications) | 2 (2)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 2 (4)
Tooth fracture (Injury, poisoning and procedural complications) | 2 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Heat exhaustion (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (2)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 1 (1)
Skeletal injury (Injury, poisoning and procedural complications) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (2)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Tooth injury (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Weight decreased (Investigations) | 30 (32)
Electrocardiogram abnormal (Investigations) | 6 (6)
Blood cholesterol increased (Investigations) | 3 (3)
Weight increased (Investigations) | 3 (3)
Blood potassium increased (Investigations) | 2 (3)
Creatinine renal clearance decreased (Investigations) | 2 (2)
Prostatic specific antigen increased (Investigations) | 2 (2)
Albumin globulin ratio increased (Investigations) | 1 (1)
Antibiotic resistant Staphylococcus test positive (Investigations) | 1 (1)
Blood calcium decreased (Investigations) | 1 (1)
Blood creatinine decreased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Body temperature increased (Investigations) | 1 (1)
Creatinine renal clearance abnormal (Investigations) | 1 (1)
Electrocardiogram ST-T change (Investigations) | 1 (1)
Electrocardiogram T wave abnormal (Investigations) | 1 (1)
Globulins increased (Investigations) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 1 (1)
Heart rate abnormal (Investigations) | 1 (1)
Occult blood positive (Investigations) | 1 (1)
Protein total increased (Investigations) | 1 (1)
Smear cervix abnormal (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (12)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Iron deficiency (Metabolism and nutrition disorders) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Magnesium deficiency (Metabolism and nutrition disorders) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Water intoxication (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Arthraglia (Musculoskeletal and connective tissue disorders) | 3 (4)
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Ostenopenia (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chorea (Nervous system disorders) | 18 (18)
Headache (Nervous system disorders) | 12 (20)
Dizziness (Nervous system disorders) | 7 (8)
Amnesia (Nervous system disorders) | 4 (4)
Somnolence (Nervous system disorders) | 4 (6)
Balance disorder (Nervous system disorders) | 3 (3)
Dysarthria (Nervous system disorders) | 3 (3)
Syncope (Nervous system disorders) | 3 (4)
Speech disorder (Nervous system disorders) | 2 (2)
Tongue biting (Nervous system disorders) | 2 (2)
Bradykinesia (Nervous system disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (2)
Dizziness postural (Nervous system disorders) | 1 (1)
Dystonia (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (8)
Paraesthesia (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Sensory loss (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 27 (29)
Insomnia (Psychiatric disorders) | 24 (28)
Depression (Psychiatric disorders) | 20 (27)
Suicidal ideation (Psychiatric disorders) | 6 (6)
Apathy (Psychiatric disorders) | 5 (5)
Agitation (Psychiatric disorders) | 4 (4)
Anger (Psychiatric disorders) | 3 (3)
Panic attack (Psychiatric disorders) | 3 (3)
Adjustment disorder (Psychiatric disorders) | 2 (2)
Bruxism (Psychiatric disorders) | 2 (4)
Delusion (Psychiatric disorders) | 2 (2)
Depressed mood (Psychiatric disorders) | 2 (3)
Obsessive-compulsive disorder (Psychiatric disorders) | 2 (2)
Paranoia (Psychiatric disorders) | 2 (2)
Alcohol abuse (Psychiatric disorders) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1)
Anhedonia (Psychiatric disorders) | 1 (1)
Bradyphrenia (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Depressive symptom (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Hypomania (Psychiatric disorders) | 1 (1)
Inappropriate affect (Psychiatric disorders) | 1 (2)
Initial insomnia (Psychiatric disorders) | 1 (1)
Nightmare (Psychiatric disorders) | 1 (1)
Obsessive thoughts (Psychiatric disorders) | 1 (1)
Perseveration (Psychiatric disorders) | 1 (1)
Pressure of speech (Psychiatric disorders) | 1 (1)
Rapid eye movements sleep abnormal (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)
Tachyphrenia (Psychiatric disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 9 (10)
Hypertonic bladder (Renal and urinary disorders) | 7 (7)
Pollakiuria (Renal and urinary disorders) | 4 (4)
Dysuria (Renal and urinary disorders) | 3 (3)
Nephrolithiasis (Renal and urinary disorders) | 3 (3)
Michurition urgency (Renal and urinary disorders) | 2 (2)
Incontinence (Renal and urinary disorders) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2)
Genital rash (Reproductive system and breast disorders) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Grunting (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiroatry tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 10 (13)
Skin lesion (Skin and subcutaneous tissue disorders) | 4 (5)
Acne (Skin and subcutaneous tissue disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Livedo reticularis (Skin and subcutaneous tissue disorders) | 2 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (2)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Generalised erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Scar (Skin and subcutaneous tissue disorders) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1)
Immobilisation prolonged (Social circumstances) | 1 (1)
Hypertension (Vascular disorders) | 4 (4)
Hot flush (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Peripheral coldness (Vascular disorders) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 1 (1)
Tooth infection (Infections and infestations) | 4 (4)

LIMITATIONS AND CAVEATS:
The study was stopped at Sponsor discretion/request; last patient last visit was 5 Jan 2018.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed. Data and results owned by Sponsor. Results can be used by institution for (a) internal non-commercial research, education and patient care, and (b) as required under applicable laws and regulations. Other uses require prior written consent of Sponsor.

DOCUMENTS (2):
  • Study Protocol (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/29/NCT01306929/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/29/NCT01306929/SAP_001.pdf